CLINICAL TRIAL: NCT00537342
Title: Prospective, Randomised, Double Blind, Placebo Controlled Study of Treatment With Sublingual Immunotherapy of Depigmented and Polymerised Allergen Extract of O. Europaea in Two Groups of Patients With Allergic Rhinitis /Rhinoconjunctivitis
Brief Title: Immunotherapy With Depigmented and Polymerized Allergen Extract of Olea Europaea (GPIT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratorios Leti, S.L. (Industry)
Responsible Party: Mª José Gómez, Laboratorios LETI S.L.Unipersonal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006-001130-41; 6018-PG-OSL-142 (Other: Sponsor protocol number)
Record Dates: First submitted 2007-09-28; First posted 2007-10-01 (Estimated); Last update posted 2010-12-17 (Estimated); Status verified 2010-12

CONDITIONS: Allergy; Rhinoconjunctivitis
Keywords: Immunotherapy; Allergoid; Depigmented; Polymerized; Allergen-extract; Rhinoconjunctivitis
MeSH Terms: conditions — Hypersensitivity | interventions — Immunotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Biological Vaccine
  Interventions: Biological: Immunotherapy with modified extract of O. europaea pollen
- B (Placebo Comparator)
  Interventions: Biological: Immunotherapy with modified extract of O. europaea pollen

INTERVENTIONS:
Biological: Immunotherapy with modified extract of O. europaea pollen — Sublingual (2 drops daily during 2 months)

SUMMARY:
The objective of this trial is to evaluate the clinical effectiveness of the administration of a depigmented and polymerized allergen extract of Olea europaea in the rhinitis or allergic rhinoconjunctivitis

DETAILED DESCRIPTION:
Immunotherapy is a specific treatment for allergic diseases. Unlike conventional pharmacological treatment, immunotherapy is the only treatment that could modify the natural course of allergic disease. This is a prospective double-blind placebo controlled study with two arms of treatment: placebo and active.

ELIGIBILITY:
Inclusion Criteria:

* Positive suggestive clinical history of allergic seasonal rhinitis or rhinoconjunctivitis
* Patients of both gender > 18 years old
* Positive prick test results using non modified Olea europaea allergen extract (wheal size > 3mm2)
* Specific IgE to Olea europaea
* Written informed consent

Exclusion Criteria:

* Use of immunotherapy during the last four years.
* Any contraindication for the use of immunotherapy in accordance with European Allergy and Clinical Immunology Immunotherapy Subcommittee criteria:
* Treatment with ß-blockers
* Coexistence of immunopathological diseases (e.g. of the liver, kidney, the nervous system, thyroid gland, rheumatic diseases) in which autoimmune mechanisms play a role
* Patients suffering from immune deficiencies
* Patients with serious psychiatric / psychological disturbances
* In addition, the following was considered as exclusion criteria:
* Pregnant or/ in lactation patients
* Patients aspirin intolerance

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2007-10; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Symptom score | 1 year

SECONDARY OUTCOMES:
Dose-response skin prick-test | 1 year
Medication score | 1 year
Rhinoconjunctivitis quality of life questionnaire | 1 year
Analogical visual scale | 1 year
Serology | 1 year
Record of adverse events | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Juan Luis Anguita, MD, Principal Investigator
Locations (1):
- Hospital Universitatio Ciudad de Jaén, Jaén, Jaén, Spain